CLINICAL TRIAL: NCT07351045
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Once-Weekly RO7795068 Administered to Participants With Obesity or Overweight Without Type 2 Diabetes
Brief Title: A Clinical Study to Evaluate the Effects of RO7795068 in Participants With Obesity or Overweight Without Type 2 Diabetes
Acronym: Enith1
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WC45725; 2025-523104-71-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo
- Arm 2: RO7795068 Dosing Regimen 1 (Experimental)
  Interventions: Combination Product: RO7795068
- Arm 3: RO7795068 Dosing Regimen 2 (Experimental)
  Interventions: Combination Product: RO7795068
- Arm 4: RO7795068 Dosing Regimen 3 (Experimental)
  Interventions: Combination Product: RO7795068

INTERVENTIONS:
Combination Product: Placebo — Placebo will be volume-matched and administered once weekly using an integrated drug-device combination product.
  Arms: Arm 1: Placebo
Combination Product: RO7795068 — RO7795068 will be administered once weekly at the randomized dosing regimen using an integrated drug-device combination product.
  Other Names: CT-388; RG6640
  Arms: Arm 2: RO7795068 Dosing Regimen 1; Arm 3: RO7795068 Dosing Regimen 2; Arm 4: RO7795068 Dosing Regimen 3

SUMMARY:
The purpose of this study is to assess the efficacy and safety of RO7795068, a dual glucagon like peptide-1 (GLP-1)/glucose-dependent insulinotropic polypeptide (GIP) receptor agonist (RA), at multiple doses compared with placebo for weight management in participants without Type 2 diabetes mellitus (T2DM) who have obesity or overweight with at least one weight-related comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at screening:

  1. Body mass index (BMI) greater than or equal to (≥)30.0 kg/m^2; or
  2. BMI ≥27.0 kg/m^2 and <30.0 kg/m^2 with at least one weight-related comorbidity, such as prediabetes, hypertension, dyslipidemia, diagnosis of obstructive sleep apnea, or weight-related cardiovascular disease
* History of ≥1 self-reported unsuccessful diet/exercise effort to lose body weight
* Ability and willingness to self-administer the study drug (or receive an injection from a trained individual if visually impaired or with physical limitations)

Exclusion Criteria:

* History of Type 1 diabetes mellitus (T1DM) or T2DM, or history of ketoacidosis or hyperosmolar state/coma. Prior, but not current, diagnosis of gestational diabetes is allowed if no history of diabetes is recorded since.
* Self-reported change in body weight >5 kg within 3 months prior to screening
* Obesity induced by other endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., melanocortin 4 receptor deficiency or Prader-Willi syndrome)
* Prior or planned surgical treatment for obesity. Liposuction or abdominoplasty if performed more than 1 year prior to screening is allowed.
* Known clinically significant gastric emptying abnormality (e.g., severe gastroparesis or gastric outlet obstruction)
* History of acute or chronic pancreatitis or clinically significant gallbladder disease. History of acute pancreatitis caused by gallstones or clinically significant gallbladder disease is allowed if the participant had a cholecystectomy to resolve the problem at least 3 months prior to screening.
* Poorly controlled hypertension at screening
* Any of the following cardiovascular conditions within 3 months prior to screening: Acute myocardial infarction; Cerebrovascular accident (stroke)/transient ischemic attack; Unstable angina; Hospitalization due to congestive heart failure.
* Have a history of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder (e.g., schizophrenia, bipolar disorder, or other serious mood or anxiety disorder). Participants with MDD or generalized anxiety disorder whose disease state is considered stable within 1 year prior to screening and expected to remain stable throughout the course of the study, in the opinion of the investigator, are allowed provided that they are not receiving prohibited medication.
* Treatment with any approved or investigational GLP-1-RA-based therapy (e.g., GLP-1 receptor mono agonist, GLP-1/GIP receptor dual agonist, GLP-1/GIP/Gluc receptor triple agonist) within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-08-07 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Percent (%) Change from Baseline in Body Weight at Week 72 | Baseline through Week 72

SECONDARY OUTCOMES:
Percentage of Participants Achieving ≥5% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥10% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥15% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥20% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Percentage of Participants Achieving ≥25% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Change from Baseline in Body Weight (kg) at Week 72 | Baseline through Week 72
Change from Baseline in Waist Circumference (cm) at Week 72 | Baseline through Week 72
Change from Baseline in Fasting Glucose at Week 72 | Baseline through Week 72
Change from Baseline in Fasting Insulin at Week 72 | Baseline through Week 72
Change from Baseline in Low-Density Lipoprotein (LDL) Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in High-Density Lipoprotein (HDL) Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Triglyceride at Week 72 | Baseline through Week 72
Change from Baseline in Systolic Blood Pressure at Week 72 | Baseline through Week 72
Change from Baseline in the Physical Functioning Domain Score of the Short Form (36) Health Survey Version 2 (SF-36v2) Acute Form at Week 72 | Baseline through Week 72
Change from Baseline in Physical Functioning Composite Score of the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQoL-Lite-CT) Questionnaire at Week 72 | Baseline through Week 72
Change from Baseline in Waist-to-Hip Ratio at Week 72 | Baseline through Week 72
Change from Baseline in Waist-to-Height Ratio at Week 72 | Baseline through Week 72
Percentage of Participants Achieving Normoglycemia (HbA1c <5.7%) at Week 72 | Baseline and Week 72
Change from Baseline in Subscale Scores of the Control of Eating Questionnaire (CoEQ) at Week 72 | Baseline through Week 72
Change from Baseline in Symptoms and Impact of Urinary Incontinence as Assessed by the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) at Week 72 | Baseline through Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the Patient Global Impression of Change (PGI-C) Urinary Incontinence Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the Patient Global Impression of Severity (PGI-S) Urinary Incontinence Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the PGI-C Physical Functioning Questionnaire at Week 72 | Baseline and Week 72
Percentage of Participants Experiencing No Change, Improvement, or Worsening on the PGI-S Physical Functioning Questionnaire at Week 72 | Baseline and Week 72
Change from Baseline in Health Related Quality of Life (HRQoL) as Assessed by the SF-36v2 Acute Form Domain Scores and Component Summary Scores at Week 72 | Baseline through Week 72
Change from Baseline in HRQoL as Assessed by the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQoL-Lite-CT) Questionnaire Domain Scores and Total Score at Week 72 | Baseline through Week 72
Change from Baseline in Non-HDL Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Total Cholesterol at Week 72 | Baseline through Week 72
Change from Baseline in Free Fatty Acids at Week 72 | Baseline through Week 72
Change from Baseline in Diastolic Blood Pressure at Week 72 | Baseline through Week 72
Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) at Week 72 | Baseline through Week 72
Percentage of Participants Achieving ≥30% Body Weight Loss from Baseline at Week 72 | Baseline and Week 72
Change from Baseline in Body Mass Index (BMI) at Week 72 | Baseline through Week 72
Percent (%) Change from Baseline in Body Weight by Obesity Class at Week 72 | Baseline through Week 72
Time to Achieve ≥5%, ≥10%, ≥15%, ≥20%, ≥25%, ≥30% Body Weight Loss from Baseline Through Week 72 | From Baseline through Week 72
Change from Baseline in Total Lean Tissue Volume (Litres) at Week 72, as Assessed by Magnetic Resonance Imaging (MRI) | Baseline through Week 72
Percent (%) Change from Baseline in Total Lean Tissue Volume at Week 72, as Assessed by MRI | Baseline through Week 72
Change from Baseline in Total Adipose Tissue Volume (Litres) at Week 72, as Assessed by MRI | Baseline through Week 72
Percent (%) Change from Baseline in Total Adipose Tissue Volume at Week 72, as Assessed by MRI | Baseline through Week 72
Incidence and Severity of Adverse Events, with Severity Determined According to Mild/Moderate/Severe Criteria | Baseline through Week 72
Change from Baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) Score Through Week 72 | Baseline through Week 72
Change from Baseline in the Patient Health Questionnaire-9 (PHQ-9) Score Through Week 72 | Baseline through Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing